CLINICAL TRIAL: NCT03945318
Title: A Phase 1/2, Multicenter Trial to Investigate the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of BION-1301 in Healthy Volunteers and Adults With IgA Nephropathy
Brief Title: Safety and Tolerability of BION-1301 in Healthy Volunteers and Adults With IgA Nephropathy (IgAN)
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CFUB523A12103; 2018-003360-31 (EudraCT Number); NCT04684745 (obsolete NCT alias)
Record Dates: First submitted 2019-04-21; First posted 2019-05-10 (Actual); Last update posted 2025-04-13 (Actual); Status verified 2025-04

CONDITIONS: IgA Nephropathy
MeSH Terms: conditions — Glomerulonephritis, IGA

STUDY DESIGN:
Intervention Model Description: Part 1 (SAD-HV) is a randomized, placebo-controlled single ascending dose design in HVs. Part 2 (MAD-HV): is a randomized, placebo-controlled multiple ascending dose design in HVs. Part 3 (MD-IgAN) is an open-label multiple dose design in participants with IgAN. Part 4 (IgAN) is open-label retreatment for Part 3 participants.
Who Masked: Participant, Care Provider, Investigator
Masking Description: Parts 1 and 2 will be performed in a double-blind manner, for clinical research personnel interacting with study participants. An unblinded pharmacist will prepare the doses of investigational study drugs.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (6):
- Part 1: BION-1301 (Experimental): Up to 5 cohorts with single ascending doses of BION-1301 administered by intravenous (IV) infusion.
  Interventions: Drug: BION-1301 Single Dose
- Part 1: Placebo (Placebo Comparator): Participants will receive a single dose of placebo administered by IV infusion.
  Interventions: Drug: Placebo Single Dose
- Part 2: BION-1301 (Experimental): Up to 4 cohorts with multiple doses of BION-1301 administered by intravenous (IV) infusion.
  Interventions: Drug: BION-1301 Multiple Doses
- Part 2: Placebo (Placebo Comparator): Participants will receive placebo by IV infusion.
  Interventions: Drug: Placebo Multiple Doses
- Part 3: BION-1301 (Experimental): Two cohorts of participants will receive multiple doses of BION-1301 by IV infusion (Cohort 1) or SC injection (Cohort 2) at 600mg/biweekly.
  Interventions: Drug: BION-1301 Multiple Doses
- Part 4 Retreatment: BION-1301 (Experimental): Eligible participants from Part 3 may enroll in Part 4 due to disease progression or by choice for optional retreatment and receive SC injection at 600mg/biweekly.
  Interventions: Drug: BION-1301 Single Dose

INTERVENTIONS:
Drug: BION-1301 Single Dose — A solution for IV infusion administered as a single dose.
  Arms: Part 1: BION-1301
Drug: Placebo Single Dose — A solution by IV infusion administered as a single dose.
  Arms: Part 1: Placebo
Drug: BION-1301 Multiple Doses — A solution for IV infusion or SC injections (Part 3 only) administered as multiple doses.
  Arms: Part 2: BION-1301; Part 3: BION-1301
Drug: Placebo Multiple Doses — A solution by IV infusion administered as multiple doses.
  Arms: Part 2: Placebo
Drug: BION-1301 Single Dose — SC injection administration as a single dose using vials or pre-filled syringes (PFS) (Part 4 only).
  Arms: Part 4 Retreatment: BION-1301

SUMMARY:
Multicenter study designed to evaluate the safety, tolerability, pharmacokinetics (PK), and pharmacodynamics (PD) of BION-1301 in healthy volunteers and adults with IgA Nephropathy (IgAN).

DETAILED DESCRIPTION:
This is a Phase 1/2 study of BION-1301, a first-in-class humanized IgG4 anti-a proliferation-inducing ligand (APRIL) monoclonal antibody.

The study will be conducted in three parts. Part 1: double-blind, randomized, placebo-controlled, single ascending dose (SAD) in healthy volunteers (HVs). Part 2: double-blind, randomized, placebo-controlled multiple ascending dose (MAD) in HVs. Part 3: Open-label, multiple dose (MD) in participants with IgAN. Part 4: Retreatment period

Parts 1 and 2 have been completed. Part 3 enrollment is complete. Part 4 enrollment is open for eligible participants from Part 3.

The study will enroll up to 40 participants with IgAN.

ELIGIBILITY:
Inclusion Criteria for Healthy Volunteers:

1. Healthy male or female volunteers, 18 to 55 years old
2. Females must be of non-childbearing potential
3. Males must agree to follow the protocol-specified contraception guidance
4. Body mass index (BMI) between 18 and 35 kg/m^2, with a weight of at least 50 kg
5. Non-smoker, defined as an individual who has not smoked previously and/or who has discontinued smoking or the use of nicotine/nicotine-containing products at least 3 months before Screening
6. Able to provide signed informed consent

Exclusion Criteria for Healthy Volunteers:

1. Regular consumption of alcohol within 6 months prior to Screening, or use of soft drugs (such as marijuana) within 3 months prior to Screening, or hard drugs (such as cocaine and phencyclidine) within 1 year prior to Screening and/or positive blood or urine test results for drugs of abuse or alcohol at Screening or Admission
2. Donated blood in the 3 months prior to the first dose of study drug, plasma in the 7 days prior to the first dose of study drug, or platelets in the 6 weeks prior to the first dose of study drug
3. History or evidence of a clinically significant disorder, condition, or disease that could pose a risk to subject safety or interfere with the study, or would make the subject unsuitable for participation, eg, respiratory, renal, hepatic, gastrointestinal, hematological, lymphatic, neurological, cardiovascular, or psychiatric disease
4. Female who is breastfeeding or who has a positive serum pregnancy test at Screening or a positive urine pregnancy test on Day -1

Inclusion Criteria for Adults with IgAN:

1. Male or female ≥18 years old at Screening
2. Women of child-bearing potential (WOCBP; per CTFG 2014) must agree to follow the protocol-specified contraception guidance throughout the study (from Screening through approximately 6 months after the final dose of study drug)
3. Males must agree to follow the protocol-specified contraception guidance throughout the study (from Screening through approximately 6 months after the final dose of study drug)
4. BMI between 18 and 40 kg/m^2, inclusive, at Screening with a weight of at least 50 kg
5. Diagnosis of IgAN verified by biopsy taken within the past 10 years
6. Urine protein ≥ 0.5 g/24h; OR UPCR ≥ 0.5 g/g (or ≥ 50 mg/mmol)
7. eGFR (per Chronic Kidney Disease Epidemiology Collaboration [CKD-EPI] formula) or measured GFR ≥ 30 mL/min per 1.73 m^2
8. Stable on an optimized dose of angiotensin converting enzyme (ACE) inhibitors and/or angiotensin-receptor blockers (ARBs) for at least 3 months prior to Screening or intolerant to ACE/ARB

Exclusion Criteria for Adults with IgAN:

1. Known or suspected allergy or hypersensitivity to any component of BION-1301, or history of severe hypersensitivity reaction to any monoclonal antibody
2. Donated blood in the 3 months prior to the first dose of study drug; plasma in the 7 days prior to the first dose of study drug; or platelets in the 6 weeks prior to the first dose of study drug
3. Participated in any other study in which receipt of an investigational new drug, or investigational device occurred within 28 days, or 5 half-lives (whichever is longer) of first dose of study drug in the present study
4. Secondary forms of IgAN as defined by the treating physician (eg, Henoch-Schönlein purpura patients and those with associated alcoholic cirrhosis)
5. Received systemic corticosteroid therapy (> 10 mg/day of prednisone or equivalent) or any other form of immunosuppressive therapy within 3 months prior to the first dose of study drug

PART 4 Eligibility Criteria for Re-treatment Due to Evidence of Disease Progression

(Option 1) Inclusion Criteria for Re-treatment Due to Evidence of Disease Progression

1. Completed Part 3 of the study through Week 124 and entered the 52-week follow-up period.
2. UPCR ≥ 0.5 g/g AND ≥ 30% increase from EOT (Week 124). Both proteinuria criteria must be met by a 24-hour urine assessment during the 52-week follow-up period. In addition to the scheduled assessments, investigators may order periodic FMV assessments (for example monthly) to follow a patient more closely. Based on an off-schedule FMV result, or other laboratory or clinical evidence, investigators may order an off-schedule 24-urine collection to confirm disease progression.

Exclusion Criteria for Re-treatment Due to Evidence of Disease Progression

1. Based on the Investigator's judgment, the patient would not benefit from resuming treatment with BION-1301 or there is a safety concern for the individual patient which outweighs the expected benefit from resuming treatment.
2. Received systemic corticosteroid therapy, including budesonide, for >14 days within 3 months prior to the first dose of Part 4 for the treatment of IgAN
3. Received any other form of immunosuppressive therapy such as, but not limited to mycophenolate mofetil, azathioprine, cyclosporine, tacrolimus, rituximab, cyclophosphamide, etc) within 3 months prior to the first dose of Part 4 study drug
4. Received investigational products for the treatment of IgAN, other than BIO-1301
5. Received newly approved immunosuppressive or immunomodulatory therapy for the treatment of IgAN including but not limited to other anti-APRIL therapies and iptacopan

Eligibility Criteria for Optional Re-treatment (Option 2)

Inclusion Criteria for Optional Re-treatment

1. Completed Part 3 of the study through Week 124 and completed of the 52-week follow-up period.

Exclusion Criteria for Optional Re-treatment

1. Based on the Investigator's judgment, the patient would not benefit from resuming treatment with BION-1301 or there is a safety concern for the individual patient which outweighs the expected benefit from resuming treatment.
2. Received systemic corticosteroid therapy, including budesonide, for >14 days within 3 months prior to the first dose in Part 4 for the treatment of IgAN
3. Received any other form of immunosuppressive therapy (such as, but not limited to mycophenolate mofetil, azathioprine, cyclosporine, tacrolimus, rituximab, cyclophosphamide, etc) within 3 months prior to the first dose of Part 4 study drug
4. Received investigational products for the treatment of IgAN, other than BIO-1301
5. Received newly approved immunosuppressive or immunomodulatory therapy for the treatment of IgAN including but not limited to other anti-APRIL therapies and iptacopan

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 103 (Actual)
Dates: Start 2019-04-08 (Actual); Primary Completion 2025-10-01 (Estimated); Study Completion 2026-04-13 (Estimated)

PRIMARY OUTCOMES:
Incidence of Treatment Emergent Adverse Events (TEAEs) as assessed according to the National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) | Participants followed from date of enrollment until the end of study, assessed up to 76 weeks.
Severity of TEAEs as assessed according to NCI-CTCAE | Participants followed from date of enrollment until the end of study, assessed up to 76 weeks.

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (16):
- United States (9):
  - Amicis Research Center, Northridge, California
  - Colorado Kidney Care, P.C., Denver, Colorado
  - Nephrology Associates of Central Florida, Orlando, Florida
  - Elixia Tampa, LLC, Tampa, Florida
  - New York Nephrology, Clifton Park, New York
  - Chris Sholer, P.C., Oklahoma City, Oklahoma
  - Liberty Research Center, Arlington, Texas
  - Liberty Research Center, Dallas, Texas
  - Prolato Clinical Research Center, Houston, Texas
- South Korea (5):
  - Soon Chun Hyang University Hospital Cheonan, Cheonan, Chungcheongnam-do
  - Hallym University Sacred Heart Hospital, Anyang-si, Gyeonggi-do
  - National Health Insurance Service Ilsan Hospital, Goyang-si, Gyeonggi-do
  - Hanyang University Guri Hostpital, Guri-si, Gyeonggi-do
  - Seoul National University Bundang Hospital, Seongnam-si, Gyeonggi-do
- United Kingdom (2):
  - Liverpool University Hospital NHS Foundation Trust, Liverpool, England
  - PAREXEL Early Phase Clinical Unit, London

IPD SHARING:
Plan to Share IPD: Yes
Novartis is committed to sharing with qualified external researchers, access to patient-level data and supporting clinical documents from eligible studies. These requests are reviewed and approved by an independent expert panel on the basis of scientific merit. All data provided is anonymized to respect the privacy of patients who have participated in the trial in line with applicable laws and regulations.
  This trial data is currently available according to the process described on www.clinicalstudydatarequest.com.

REFERENCES:
- [Derived] Kooienga L, Lo J, Lee EY, Kim SG, Thomas H, Workeneh B, Agha I, Song Y, Smith W, van Eenennaam H, Van Elsas A, Dulos J, Barratt J. Zigakibart demonstrates clinical safety and efficacy in a Phase 1/2 trial of healthy volunteers and patients with IgA nephropathy. Kidney Int. 2025 Sep;108(3):445-454. doi: 10.1016/j.kint.2025.05.006. Epub 2025 Jun 5. PMID 40482854